CLINICAL TRIAL: NCT03689777
Title: The Impact of Bariatric Surgery on Estimated Glomerular Filtration Rate in Chinese Obesity Patients: a Retrospective Cohort Study
Brief Title: the Related Factors of Bariatric Surgery on Glomerular Filtration Rate
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: First Affiliated Hospital of Jinan University (Other)
Responsible Party: Principal Investigator, Jingge Yang, Director of bariatric surgery, First Affiliated Hospital of Jinan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: FirstJinanU20180212
Record Dates: First submitted 2018-06-03; First posted 2018-09-28 (Actual); Last update posted 2018-09-28 (Actual); Status verified 2018-09

CONDITIONS: Bariatric Surgery; Glomerular Filtration Rate
MeSH Terms: interventions — Gastric Bypass

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Glomerular Filtration Rate (Active Comparator)
  Interventions: Procedure: sleeve gastrectomy; Procedure: gastric bypass

INTERVENTIONS:
Procedure: sleeve gastrectomy — sleeve gastrectomy
Procedure: gastric bypass — gastric bypass

SUMMARY:
Obesity and related metabolic diseases have become a chronic disease that is a threat to human health. Bariatric surgery can effectively and long-term reduce excess body weight and relieve related metabolic diseases, including type 2 diabetes. Laparoscopic gastric bypass surgery and laparoscopic sleeve gastrectomy are commonly used in bariatric surgery. Laparoscopic sleeve gastrectomy due to simple operation, good weight loss, and metabolic disease control effect, which is more widely used. However, there are several studies that show an increased chance of gastroesophageal reflux disease after laparoscopic sleeve gastrectomy. Long-term gastroesophageal reflux may lead to Barrett's esophagus or esophageal cancer. Nowadays, the cause of gastroesophageal reflux disease after sleeve gastrectomy is not clear and precautionary measures are not precise.

In this study, prospective randomized controlled trials were conducted to explore the possible causes of glomerular filtration rate after bariatric surgery and to explore ways to prevent glomerular filtration rate after the surgery

DETAILED DESCRIPTION:
With the social development and changes in the lifestyle, the incidence of obesity and type 2diabetes is rapidly increasing. In 2010, the global incidence of type 2 diabetes was 8.3% in adults, 11.6% in China and 50.1% in China. In overweight and obese people, the prevalence of type 2 diabetes also increased significantly, and the prevalence of type 2diabetes in those people with BMI> 30 reached 18.5-23%. Diabetes-induced cardiovascular and cerebrovascular diseases, renal insufficiency and other complications, seriously affecting the quality of life of the patients, endangering the safety of life, the treatment of type 2 diabetes and related complications to public health expenditure has brought tremendous pressure.

Traditional medical methods are difficult to achieve long-term and effective control of type 2 diabetes. Surgery has been shown to achieve 75-95% long-term relief of obesity in patients. Roux-en-Y gastric bypass (Roux-en-Y gastric bypass, RYGB) and laparoscopic sleeve gastrectomy are most commonly used. Among them, laparoscopic sleeve gastrectomy is relatively simple, low incidence of complications, lower operating costs, and gradually become the most important surgical methods of weight loss and metabolic disease surgery. Numerous clinical studies are shown that sleeve gastrectomy in patients with type 2 diabetes has the same therapeutic effect as gastric bypass with a complete remission rate of 70-90% for T2DM.

For the choice of surgical approach, numerous studies have shown that BMI ≧ 45, the general choice of gastric bypass surgery, BMI <45, you can choose sleeve gastrectomy. The remission rate for T2DM, sleeve gastrectomy has a good result for young patients with shorter duration. In our country, the BMI less than 45 is majorities.

ELIGIBILITY:
Inclusion Criteria:

-For the choice of surgical approach, numerous studies have shown that BMI ≧ 45, the general choice of gastric bypass surgery, BMI <45, you can choose sleeve gastrectomy. The remission rate for T2DM, sleeve gastrectomy has a good result for young patients with shorter duration. In our country, the BMI less than 45 is majorities.

Exclusion Criteria:

-BMI<27.5

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1000 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
preoperative of glomerular filtration rate | Preoperative
  Glomerular Filtration Rate in ml/min
Postoperative of glomerular filtration rate at 3 months | 3 months
  Glomerular Filtration Rate in ml/min
Postoperative of glomerular filtration rate at 6 months | 6 months
  Glomerular Filtration Rate in ml/min
Postoperative of glomerular filtration rate at 1 year | 1 year
  Glomerular Filtration Rate in ml/min

CONTACTS AND LOCATIONS:
Locations (1):
- The frist affiliated hospital of Jinan University, Guangzhou, Guangdong, China